CLINICAL TRIAL: NCT00321919
Title: A Randomized, Open-label Study of the Effect of NeoRecormon on Reduction of Cardiovascular Risk in Patients With Chronic Renal Anemia Who Are Not on Renal Replacement Therapy.
Brief Title: A Study of Treatment With NeoRecormon (Epoetin Beta) in Patients With Chronic Renal Anemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BA16169
Record Dates: First submitted 2006-05-03; First posted 2006-05-04 (Estimated); Results first posted 2016-05-25 (Estimated); Last update posted 2016-06-29 (Estimated); Status verified 2016-05

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — epoetin beta

ARMS (2):
- Early Epoetin Beta Therapy (Experimental): Participants received immediate epoetin beta therapy starting at 2000 IU, subcutaneously once weekly up to four years to reach a target Hb level of 13-15 g/dL; with an individual Hb increase of at least 2 g/dL within approximately 3 months.
  Interventions: Drug: epoetin beta [NeoRecormon]
- Late Epoetin Beta Therapy (Active Comparator): Participants received epoetin beta treatment starting at 2000 IU, subcutaneously once weekly up to four years only when a decline in Hb levels to <10.5 g/dL had occurred in order to reach a target Hb of 10.5-11.5 g/dL.
  Interventions: Drug: epoetin beta [NeoRecormon]

INTERVENTIONS:
Drug: epoetin beta [NeoRecormon] — Participants in the early treatment group immediately started epoetin beta treatment to reach a target Hb level of 13-15 g/dL at the end of the correction phase.
  Arms: Early Epoetin Beta Therapy
Drug: epoetin beta [NeoRecormon] — Participants in the late treatment Group started epoetin beta treatment once a decline in Hb level to <10.5 g/dL had occurred.
  Arms: Late Epoetin Beta Therapy

SUMMARY:
This study will evaluate whether anemia prevention with NeoRecormon has an additional impact on reducing cardiovascular risk over conventional anemia treatment in patients mostly with stage IV chronic kidney disease and renal anemia. The anticipated time on study treatment is 2+ years and the target sample size is 500+ individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients >=18 years of age;
* chronic renal anemia;
* not receiving renal replacement therapy.

Exclusion Criteria:

* women who are pregnant or lactating;
* previous treatment with erythropoietin or other erythropoietic substance;
* blood transfusion within the last 3 months;
* need for dialysis expected in the next 6 months;
* administration of another investigational drug within 30 days preceding study start, or during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 605 (Actual)
Dates: Start 2000-07; Primary Completion 2004-10 (Actual); Study Completion 2004-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (86):
- Austria (2):
  - Linz
  - Sankt Pölten
- Belgium (2):
  - Brussels
  - Edegem
- Czechia (4):
  - Brno
  - Havířov
  - Olomouc
  - Ostrava
- Denmark (4):
  - Fredericia
  - Herlev
  - Holbæk
  - Roskilde
- Finland (2):
  - Jyväskylä
  - Tampere
- France (11):
  - Amiens
  - Angoulême
  - Bordeaux
  - Boulogne
  - Colmar
  - Lyon
  - Montpellier
  - Paris
  - Saint-Brieuc
  - Troyes
  - Vandœuvre-lès-Nancy
- Germany (3):
  - Berlin
  - Villingen-Schwenningen
  - Würzburg
- Greece (3):
  - Athens
  - Thessaloniki
  - Véria
- Hong Kong, Hong Kong
- Dublin, Ireland
- Italy (13):
  - Bologna
  - Busto Arsizio
  - Cagliari
  - Cinisello Balsamo
  - Lecco
  - Napoli
  - Padua
  - Parma
  - Pavia
  - Roma
  - San Giovanni Rotondo
  - Trieste
  - Vimercate
- Mexico (2):
  - Cuernavaca
  - Tijuana
- Oslo, Norway
- Poland (4):
  - Gdansk
  - Kielce
  - Krakow
  - Wroclaw
- Portugal (4):
  - Almada
  - Carnaxide
  - Lisbon
  - Porto
- Russia (2):
  - Moscow
  - Saint Petersburg
- Spain (4):
  - Barcelona
  - Las Palmas de Gran Canaria
  - Madrid
  - Valencia
- Sweden (8):
  - Borås
  - Helsingborg
  - Jönköping
  - Karlstad
  - Norrköping
  - Örebro
  - Stockholm
  - Sundsvall
- Taiwan (4):
  - Taichung
  - Tainan
  - Taipei
  - Taoyuan District
- Thailand (2):
  - Bangkok
  - Chiang Mai
- Turkey (Türkiye) (3):
  - Ankara
  - Istanbul
  - Izmir
- United Kingdom (6):
  - Belfast
  - London
  - Newcastle upon Tyne
  - Salford
  - Southampton
  - Surrey

REFERENCES:
- [Derived] Chung EY, Palmer SC, Saglimbene VM, Craig JC, Tonelli M, Strippoli GF. Erythropoiesis-stimulating agents for anaemia in adults with chronic kidney disease: a network meta-analysis. Cochrane Database Syst Rev. 2023 Feb 13;2(2):CD010590. doi: 10.1002/14651858.CD010590.pub3. PMID 36791280
- [Derived] Locatelli F, Eckardt KU, Macdougall IC, Tsakiris D, Clyne N, Burger HU, Scherhag A, Drueke TB; Cardiovascular Risk Reduction in Early Anaemia Trial with Epoetin Beta investigators and coordinators. Value of N-terminal brain natriuretic peptide as a prognostic marker in patients with CKD: results from the CREATE study. Curr Med Res Opin. 2010 Nov;26(11):2543-52. doi: 10.1185/03007995.2010.516237. Epub 2010 Sep 17. PMID 20849244
- [Derived] Drueke TB, Locatelli F, Clyne N, Eckardt KU, Macdougall IC, Tsakiris D, Burger HU, Scherhag A; CREATE Investigators. Normalization of hemoglobin level in patients with chronic kidney disease and anemia. N Engl J Med. 2006 Nov 16;355(20):2071-84. doi: 10.1056/NEJMoa062276. PMID 17108342

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted from 26 July 2000 to 13 December 2004 at 94 centers in 21 countries.
Pre-assignment Details: Of the 605 participants, 603 started the study; 2 were withdrawn from the study due to non-compliance with good clinical practice and were excluded from the analysis.
Groups:
- Early Epoetin Beta Therapy: Participants received immediate epoetin beta therapy starting at 2000 IU, subcutaneously once weekly up to four years to reach a target Hemoglobin (Hb) level of 13-15 gram/decilitre (g/dL) with an individual Hb increase of at least 2 g/dL within approximately 3 months.
- Late Epoetin Beta Therapy: Participants received epoetin beta treatment starting at 2000 IU, subcutaneously once weekly up to four years only when a decline in Hb levels to <10.5 g/dL has occurred in order to reach a target Hb of 10.5-11.5 g/dL.
Period: Overall Study
Arm/Group | Early Epoetin Beta Therapy | Late Epoetin Beta Therapy
Started | 301 | 302
Completed | 226 | 250
Not Completed | 75 | 52
Not completed — Adverse Event | 17 | 10
Not completed — Death | 21 | 17
Not completed — Insufficient Therapeutic Response | 1 | 0
Not completed — Violation of Selection Criteria at Entry | 1 | 1
Not completed — Refused Treatment | 23 | 14
Not completed — Other Protocol Violation | 2 | 3
Not completed — Failure to Return | 3 | 1
Not completed — Other withdrawal reason | 7 | 6

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were described for the intent-to-treat (ITT) population, which included all participants randomized according to their randomized treatment group, regardless of the treatment actually received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Early Epoetin Beta Therapy | Late Epoetin Beta Therapy | Total
Number analyzed (Participants) | 301 | 302 | 603
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.3 (14.57) | 58.8 (13.73) | 59.0 (14.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 130 | 148 | 278
  Male | 171 | 154 | 325

OUTCOME MEASURES:

1. Primary Outcome: Median Time to First Cardiovascular Event
Description: The cardiovascular event was defined as any of the following: angina pectoris leading to hospitalization for at least 24 hours or prolongation of hospitalization, acute heart failure, fatal or non-fatal myocardial infarction, fatal or non-fatal stroke, sudden death, transient cerebral ischemic attack (TIA), peripheral vascular disease (amputation, necrosis), cardiac arrhythmias leading to hospitalization for at least 24 hours or prolongation of hospitalization. The time to occurrence of a cardiovascular event was determined as the time from randomization until any of the above listed events whichever occurred first. The first event per participant was used for the analysis. Only events confirmed by the Endpoint Committee were considered for analysis.
Time Frame: Up to 4 years
Population: The ITT population included all participants randomized according to their randomized treatment group, regardless of the treatment actually received.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Early Epoetin Beta Therapy | Late Epoetin Beta Therapy
Number analyzed (Participants) | 301 | 302
days | NA [NA to NA] — Data was not available due to insufficient number of participants with cardiovascular events. | NA [NA to NA] — Data was not available due to insufficient number of participants with cardiovascular events.
Statistical Analysis 1: Comparison: Early Epoetin Beta Therapy vs Late Epoetin Beta Therapy; The null hypothesis stated that there was no difference with regard to the event-free distribution of the combined endpoint of all protocol specified cardiovascular events between Early Epoetin beta therapy and Late Epoetin beta therapy groups; Test type: Superiority or Other; p = 0.2036, Regression, Cox; Risk Ratio (RR) = 0.778976, 95% CI 2-sided [0.53 to 1.14] — The Cox regression model was used to estimate the relative risk of the time to first cardiovascular event in Late Epoetin beta therapy group compared to the Early Epoetin beta therapy group

2. Secondary Outcome: Median Time to Death Due to Cardiovascular Events
Description: Time to death due to cardiovascular events is the time determined between randomization and death due to cardiovascular events.
Time Frame: Up to 4 years
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Early Epoetin Beta Therapy | Late Epoetin Beta Therapy
Number analyzed (Participants) | 301 | 302
days | NA [NA to NA] — Data was not available due to insufficient number of deaths due to cardiovascular events. | NA [NA to NA] — Data was not available due to insufficient number of deaths due to cardiovascular events.
Statistical Analysis 1: Comparison: Early Epoetin Beta Therapy vs Late Epoetin Beta Therapy; Test type: Superiority or Other; p = 0.4833, Regression, Cox; Risk Ratio (RR) = 0.744575, 95% CI 2-sided [0.33 to 1.70] — The Cox regression model was used to estimate the relative risk of an event of the time to death due to cardiovascular reasons in Late Epoetin beta therapy group compared to the Early Epoetin beta therapy group

3. Secondary Outcome: Number of Participants Who Died Due to Cardiovascular Events
Description: The cardiovascular event was defined as any of the following: angina pectoris leading to hospitalization for at least 24 hours or prolongation of hospitalization, acute heart failure, fatal or non-fatal myocardial infarction, fatal or non-fatal stroke, sudden death, transient cerebral ischemic attack (TIA), peripheral vascular disease (amputation, necrosis), cardiac arrhythmias leading to hospitalization for at least 24 hours or prolongation of hospitalization.
Time Frame: Up to 4 years
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Early Epoetin Beta Therapy | Late Epoetin Beta Therapy
Number analyzed (Participants) | 301 | 302
participants
  Total Cardiovascular Death Events | 8 | 6
  Cardiac Failure | 1 | 2
  Cardiac Failure Acute | 1 | 2
  Acute Myocardial Infarction | 1 | 1
  Angina Pectoris | 1 | 0
  Arrhythmia | 1 | 0
  Cardiac Arrest | 1 | 0
  Cardio-Respiratory Arrest | 1 | 0
  Cardiopulmonary Failure | 1 | 0
  Myocardial Infarction | 0 | 1

4. Secondary Outcome: Median Time to Death Due to All Causes
Description: Time to death due to all causes is the time determined between randomization and death due to all causes.
Time Frame: Up to 4 years
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Early Epoetin Beta Therapy | Late Epoetin Beta Therapy
Number analyzed (Participants) | 301 | 302
days | NA [NA to NA] — Data was not available due to insufficient number of deaths due to all causes. | NA [NA to NA] — Data was not available due to insufficient number of deaths due to all causes.
Statistical Analysis 1: Comparison: Early Epoetin Beta Therapy vs Late Epoetin Beta Therapy; Test type: Superiority or Other; p = 0.1391, Regression, Cox; Risk Ratio (RR) = 0.658259, 95% CI 2-sided [0.38 to 1.15] — The Cox regression model was used to estimate the relative risk of the time to death for all causes in Late Epoetin beta therapy group compared to the Early Epoetin beta therapy treatment group

5. Secondary Outcome: Number of Participants Who Died Due to All Causes
Description: Number of participants who died due to all causes are presented in table below.
Time Frame: Up to 4 years
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Early Epoetin Beta Therapy | Late Epoetin Beta Therapy
Number analyzed (Participants) | 301 | 302
participants
  Total Death Events for All-cause | 31 | 21
  Sudden Death | 4 | 2
  Cerebrovascular Accident | 2 | 2
  Cardiac Failure | 1 | 2
  Cardiac Failure Acute | 1 | 2
  Sepsis | 1 | 2
  Acute Myocardial Infarction | 1 | 1
  Bronchopneumonia | 1 | 1
  Respiratory Failure | 1 | 1
  Septic Shock | 2 | 0
  Acute Heart Failure | 1 | 0
  Acute Respiratory Failure | 0 | 1
  Angina Pectoris | 1 | 0
  Arrhythmia | 1 | 0
  Cardiac Arrest | 1 | 0
  Cardio-Respiratory Arrest | 1 | 0
  Cardiopulmonary Failure | 1 | 0
  Cerebral Infarction | 1 | 0
  Clostridial Infection | 1 | 0
  Colon Cancer Metastatic | 0 | 1
  Embolic Stroke | 1 | 0
  Intestinal Infarction | 0 | 1
  Intestinal Ischaemia | 0 | 1
  Laryngeal Cancer | 1 | 0
  Lung Neoplasm Malignant | 0 | 1
  Metastases To Lung | 1 | 0
  Metastatic Neoplasm | 1 | 0
  Myocardial Infarction | 0 | 1
  Oesophageal Carcinoma | 1 | 0
  Peripheral Vascular Disorder | 1 | 0
  Pneumonia | 0 | 1
  Pulmonary Embolism | 0 | 1
  Renal Failure | 1 | 0
  Unevaluable Event | 1 | 0
  Uraemic Encephalopathy | 1 | 0

6. Secondary Outcome: Number of Participants Experiencing Worsening of New York Heart Association (NYHA) Class (CL) of Chronic Heart Failure From Baseline (BL)
Description: The NYHA functional classification assesses the severity of symptoms of chronic heart failure and is comprised of four classes. Class I is defined as no limitation of physical activity, Class II is defined as slight limitation of physical activity, Class III is defined as marked limitation of physical activity, and Class IV is defined as unable to carry on any physical activity without discomfort. Shifts of participants from CL 0, CL I, CL II, CL III, CL IV at Baseline (Day 1) to CL 0, CL I, CL II, CL III, CL IV during the study period was determined and presented.
Time Frame: Up to 4 years
Population: The ITT population included all participants randomized according to their randomized treatment group, regardless of the treatment actually received. The "n" represents the number of participants assessed for shifts in NYHA class from baseline.
Measure: Number; unit: participants
Arm/Group | Early Epoetin Beta Therapy | Late Epoetin Beta Therapy
Number analyzed (Participants) | 167 | 149
participants
  From CL 0 (BL) to CL 0; n = 167, 149 | 49 | 42
  From CL 0 (BL) to CL I; n = 167, 149 | 7 | 4
  From CL 0 (BL) to CL II; n = 167, 149 | 7 | 7
  From CL 0 (BL) to CL III; n = 167, 149 | 2 | 1
  From CL 0 (BL) to CL IV; n = 167, 149 | 0 | 0
  From CL I (BL) to CL 0; n = 37, 43 | 1 | 0
  From CL I (BL) to CL I; n = 37, 43 | 28 | 34
  From CL I (BL) to CL II; n = 37, 43 | 5 | 4
  From CL I (BL) to CL III; n = 37, 43 | 0 | 0
  From CL I (BL) to CL IV; n = 37, 43 | 0 | 0
  From CL II (BL) to CL 0; n = 53, 44 | 0 | 0
  From CL II (BL) to CL I; n = 53, 44 | 5 | 1
  From CL II (BL) to CL II; n = 53, 44 | 39 | 37
  From CL II (BL) to CL III; n = 53, 44 | 2 | 4
  From CL II (BL) to CL IV; n = 53, 44 | 0 | 0
  From CL III (BL) to CL 0; n = 0, 0 | 0 | 0
  From CL III (BL)to CL I; n = 0, 0 | 0 | 0
  From CL III (BL)to CL II; n = 0, 0 | 0 | 0
  From CL III (BL)to CL III; n = 0, 0 | 0 | 0
  From CL III (BL)to CL IV; n = 0, 0 | 0 | 0
  From CL IV (BL)to CL 0; n = 0, 0 | 0 | 0
  From CL IV (BL)to CL I; n = 0, 0 | 0 | 0
  From CL IV (BL)to CL II; n = 0, 0 | 0 | 0
  From CL IV (BL)to CL III; n = 0, 0 | 0 | 0
  From CL IV (BL)to CL IV; n = 0, 0 | 0 | 0

7. Secondary Outcome: Median Time to First Cardiovascular Intervention
Description: Time to first cardiovascular intervention is the time between randomization and first intervention determined for all cardiovascular interventions after randomization. Cardiovascular interventions considered were: angioplasty with or without stents/atherectomy, coronary artery bypass surgery, cardioverter defibrillator (CD) cardioversion/defibrillation, temporary pacemaker, permanent pacemaker and implantable cardioverter defibrillator (ICD) implantation.
Time Frame: Up to 4 years
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Early Epoetin Beta Therapy | Late Epoetin Beta Therapy
Number analyzed (Participants) | 301 | 302
days | NA [NA to NA] — Data was not available due to insufficient number of cardiovascular interventions. | NA [NA to NA] — Data was not available due to insufficient number of cardiovascular interventions.
Statistical Analysis 1: Comparison: Early Epoetin Beta Therapy vs Late Epoetin Beta Therapy; Test type: Superiority or Other; p = 0.4985, Regression, Cox; Risk Ratio (RR) = 0.804594, 95% CI 2-sided [0.43 to 1.51] — The Cox regression model was used to estimate the relative risk of time to first cardiovascular intervention in Late Epoetin beta therapy group compared to the Early Epoetin beta therapy group

8. Secondary Outcome: Total Number of Cardiovascular Intervention
Description: Cardiovascular intervention was defined by a clinical review of all concomitant treatments. The cardiovascular interventions considered were: angioplasty with or without stents/atherectomy, coronary artery bypass surgery, cardioverter defibrillator (CD) cardioversion/defibrillation, temporary pacemaker, permanent pacemaker and implantable cardioverter defibrillator (ICD) implantation. The total number of cardiovascular intervention was determined and presented by each cohort.
Time Frame: Up to 4 years
Population: as for outcome 1
Measure: Number; unit: number of cardiovascular intervention
Arm/Group | Early Epoetin Beta Therapy | Late Epoetin Beta Therapy
Number analyzed (Participants) | 301 | 302
number of cardiovascular intervention | 21 | 18

9. Secondary Outcome: Median Time to First Hospitalization Due to Cardiovascular Events
Description: Time to first hospitalization due to cardiovascular events is defined as the time determined between randomization and first hospitalization due to cardiovascular events.
Time Frame: Up to 4 years
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Early Epoetin Beta Therapy | Late Epoetin Beta Therapy
Number analyzed (Participants) | 301 | 302
days | NA [NA to NA] — Data was not available due to insufficient number of hospitalizations due to cardiovascular events. | NA [NA to NA] — Data was not available due to insufficient number of hospitalizations due to cardiovascular events.
Statistical Analysis 1: Comparison: Early Epoetin Beta Therapy vs Late Epoetin Beta Therapy; Test type: Superiority or Other; p = 0.3419, Regression, Cox; Risk Ratio (RR) = 0.82046, 95% CI 2-sided [0.55 to 1.23] — The Cox regression model was used to estimate the relative risk of the time to first hospitalization for cardiovascular reasons in Late Epoetin beta therapy group compared to the Early Epoetin beta therapy group

10. Secondary Outcome: Duration of Hospitalization for Cardiovascular Events
Description: The duration of hospitalization was the total number of days that a participant was hospitalized due to cardiovascular events. Participants with no hospitalization were excluded from analysis.
Time Frame: Up to 4 years
Population: The ITT population included all participants randomized according to their randomized treatment group, regardless of the treatment actually received. Data for the participants present at the time of assessment was used for analysis.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Early Epoetin Beta Therapy | Late Epoetin Beta Therapy
Number analyzed (Participants) | 171 | 161
days | 33.0 (42.0) | 28.2 (33.7)

11. Secondary Outcome: Mean Change From Baseline in Left Ventricular Mass Index (LVMI)
Description: LVMI is determined by echocardiogram. LVMI indexed to body surface area (gram/square meter) estimated by LV cavity dimension and wall thickness at end-diastole. The change was calculated as week value minus baseline value.
Time Frame: Baseline, Week 12, Week 24, Week 36, and Week 48
Population: The ITT population included all participants randomized according to their randomized treatment group, regardless of the treatment actually received. The "n" represents the number of participants assessed for LVMI at Baseline, Week 12, Week 24, Week 36, and Week 48.
Measure: Mean (Standard Deviation); unit: gram/square meter
Arm/Group | Early Epoetin Beta Therapy | Late Epoetin Beta Therapy
Number analyzed (Participants) | 219 | 232
gram/square meter
  LVMI, Baseline; n = 219, 232 | 120.32 (35.03) | 117.97 (34.34)
  LVMI, Week 12; n = 171, 186 | -5.06 (24.81) | -2.87 (25.16)
  LVMI, Week 24; n = 136, 146 | -6.58 (26.94) | -7.59 (25.59)
  LVMI, Week 36; n = 74, 81 | -1.30 (36.04) | -7.53 (34.37)
  LVMI, Week 48; n = 2, 11 | 2.00 (2.83) | -27.27 (29.47)

12. Secondary Outcome: Mean Change From Baseline in Left Ventricular Ejection Fraction (LVEF) and Fractional Myocardial Shortening (FS)
Description: LVEF is a marker of left ventricular systolic function and determined by echocardiogram. It is expressed as the ratio of left ventricular stroke volume (LVSV) to left ventricular end-diastolic volume (LVEDV), and is measured as a percentage. FS is used as an estimate of myocardial contractility and determined by echocardiogram and measures as a percentage. The change for LVEF and FS was calculated as Week value minus baseline value.
Time Frame: Baseline, Week 12, Week 24, Week 36, and Week 48
Population: The ITT population included all participants randomized according to their randomized treatment group, regardless of the treatment actually received. The "n" represents the number of participants assessed for LVEF and FS at Baseline, Week 12, Week 24, Week 36, and Week 48.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Early Epoetin Beta Therapy | Late Epoetin Beta Therapy
Number analyzed (Participants) | 219 | 233
percentage
  LVEF, Baseline; n = 219, 233 | 81.31 (7.24) | 81.95 (7.75)
  LVEF, Week 12; n = 170, 186 | -0.08 (7.32) | 0.08 (7.34)
  LVEF, Week 24; n = 135, 147 | -0.47 (6.82) | -0.23 (7.01)
  LVEF, Week 36; n = 74, 81 | -0.61 (8.61) | 0.24 (6.75)
  LVEF, Week 48; n = 2,11 | -0.46 (2.92) | 2.80 (8.12)
  FS, Baseline; n = 219, 232 | 43.67 (7.12) | 44.67 (7.86)
  FS, Week 12; n = 196, 212 | 0.13 (6.79) | 0.08 (7.34)
  FS, Week 24; n = 174, 192 | 0.11 (7.10) | -0.19 (7.40)
  FS, Week 36; n = 98, 105 | 0.05 (8.16) | 0.70 (7.80)
  FS, Week 48; n = 4,12 | 1.00 (2.83) | 3.00 (8.58)

13. Secondary Outcome: Mean Change From Baseline in Left Ventricular Volume (LV Volume )
Description: Left Ventricular Volume is the estimated of left ventricular end-diastolic volume (LVEDv) and left ventricular end-systolic volume (LVESV) determined by Echocardiogram. The change was calculated as week value minus baseline value.
Time Frame: Baseline, Week 12, Week 24, Week 36, and Week 48
Population: The ITT population included all participants randomized according to their randomized treatment group, regardless of the treatment actually received. The "n" represents the number of participants assessed for LV Volume at Baseline, Week 12, Week 24, Week 36 and Week 48.
Measure: Mean (Standard Deviation); unit: milliliters per meter square
Arm/Group | Early Epoetin Beta Therapy | Late Epoetin Beta Therapy
Number analyzed (Participants) | 218 | 232
milliliters per meter square
  LV Volume, Baseline; n = 218, 232 | 67.73 (19.20) | 65.11 (19.24)
  LV Volume, Week 12; n = 170, 186 | -2.83 (15.90) | 3.15 (15.46)
  LV Volume, Week 24; n = 134, 146 | -0.69 (16.44) | 2.62 (18.56)
  LV Volume, Week 36; n = 72, 80 | 3.34 (24.29) | 4.05 (19.08)
  LV Volume, Week 48; n = 2, 11 | 14.48 (11.52) | 7.91 (23.37)

14. Secondary Outcome: Mean Values of Echocardiography Parameters
Description: Mean values of Echocardiography (ECHO) Parameters: Left Ventricular End Diastolic Diameter (LVEDD), Left Ventricular Posterior Wall Thickness (LVPWT), IV Septal Wall Thickness (IVSWT), LV End Systolic Diameter (LVESD), LV Relative wall thickness (LVRWT) at Baseline, Year 1, Year 2, Year 3 and Year 4 were presented.
Time Frame: Baseline, Year 1, Year 2, Year 3, and Year 4
Population: The ITT population included all participants randomized according to their randomized treatment group, regardless of the treatment actually received. The "n" represents the number of participants assessed for each echocardiography parameter at Baseline, Year 1, Year 2, Year 3 and Year 4.
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Early Epoetin Beta Therapy | Late Epoetin Beta Therapy
Number analyzed (Participants) | 219 | 233
centimeters
  LVEDD, Baseline, n = 219, 233 | 5.05 (0.67) | 4.91 (0.68)
  LVEDD, Year 1, n = 170, 186 | 4.93 (0.62) | 4.94 (0.65)
  LVEDD, Year 2, n = 135, 147 | 4.95 (0.63) | 4.93 (0.72)
  LVEDD, Year 3, n = 74, 81 | 5.09 (0.71) | 4.88 (0.59)
  LVEDD, Year 4, n = 2,11 | 5.21 (0.30) | 5.08 (0.79)
  LVPWT, Baseline, n = 219, 233 | 1.05 (0.17) | 1.05 (0.17)
  LVPWT, Year 1, n = 170, 186 | 1.02 (0.17) | 1.01 (0.16)
  LVPWT, Year 2, n= 135, 147 | 1.01 (0.13) | 0.99 (0.14)
  LVPWT, Year 3, n = 74, 81 | 1.01 (0.17) | 1.00 (0.13)
  LVPWT, Year 4, n = 2,11 | 1.08 (0.13) | 0.92 (0.16)
  IVSWT, Baseline, n = 219, 233 | 1.18 (0.24) | 1.20 (0.28)
  IVSWT, Year 1, n = 170, 186 | 1.17 (0.23) | 1.13 (0.24)
  IVSWT, Year 2, n = 135, 147 | 1.12 (0.21) | 1.11 (0.20)
  IVSWT, Year 3, n = 74, 81 | 1.14 (0.25) | 1.12 (0.22)
  IVSWT, Year 4, n = 2, 11 | 1.30 (0.05) | 1.04 (0.20)
  LVESD, Baseline, n = 219, 233 | 2.85 (0.58) | 2.74 (0.66)
  LVESD, Year 1, n = 170, 186 | 2.76 (0.56) | 2.73 (0.62)
  LVESD, Year 2, n = 135, 147 | 2.78 (0.58) | 2.75 (0.68)
  LVESD, Year 3, n = 74, 81 | 2.88 (0.75) | 2.67 (0.59)
  LVESD, Year 4, n = 2, 11 | 2.93 (0.22) | 2.84 (0.57)
  LVRWT, Baseline, n = 219, 233 | 0.42 (0.08) | 0.43 (0.09)
  LVRWT, Year 1, n = 170, 186 | 0.42 (0.08) | 0.41 (0.08)
  LVRWT, Year 2, n = 135, 147 | 0.41 (0.06) | 0.41 (0.07)
  LVRWT, Year 3, n = 74, 81 | 0.41 (0.09) | 0.42 (0.07)
  LVRWT, Year 4, n = 2, 11 | 0.41 (0.03) | 0.37 (0.07)

15. Secondary Outcome: Mean Values of Body Surface Area
Description: The body surface area (BSA) was determined by Echocardiogram. Absolute mean values of Echocardiography (ECHO) Parameter: Body surface area (BSA) at Baseline, Year 1, Year 2, Year 3 and Year 4 were calculated and presented.
Time Frame: Baseline, Year 1, Year 2, Year 3, and Year 4.
Population: The ITT population included all participants randomized according to their randomized treatment group, regardless of the treatment actually received. The "n" represents the number of participants assessed for Body surface area through echocardiogram at Baseline, Year 1, Year 2, Year 3 and Year 4.
Measure: Mean (Standard Deviation); unit: Square meter
Arm/Group | Early Epoetin Beta Therapy | Late Epoetin Beta Therapy
Number analyzed (Participants) | 287 | 290
Square meter
  BSA, Baseline, n = 287, 290 | 1.83 (0.22) | 1.79 (0.20)
  BSA, Year 1, n = 257, 261 | 1.83 (0.22) | 1.77 (0.23)
  BSA, Year 2, n = 224, 234 | 1.82 (0.21) | 1.77 (0.19)
  BSA, Year 3, n = 116, 121 | 1.82 (0.21) | 1.72 (0.19)
  BSA, Year 4, n = 4, 11 | 1.96 (0.21) | 1.76 (0.22)

16. Secondary Outcome: Mean Change From Baseline in the Scores of Each of The Eight Health Scales of Quality of Life Based on Short Form-36 (SF-36) Questionnaire
Description: The Quality of life was assessed on the basis of a change from baseline in the scores of each of the eight health scales in the SF-36 questionnaire. The SF-36 is a standardized survey evaluating 8 domains (consisting of 2 components; physical and mental) of functional health and well-being: physical and social functioning, physical and emotional role (role-physical, role-emotional) limitations, bodily pain, general health (GH), vitality, mental health. The score for a section is an average of the individual question scores, which are scaled from 0 (worst level of functioning) to 100 (100=best level of functioning). The least squares mean (LSM) change from baseline was determined by Analysis of covariance (ANCOVA) model and presented for each of the eight health scale.
Time Frame: Baseline, Year 1, and Year 2
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Early Epoetin Beta Therapy | Late Epoetin Beta Therapy
Number analyzed (Participants) | 301 | 302
units on a scale
  General Health, Year 1 | 4.1 (1.01) | -0.1 (0.99)
  General Health, Year 2 | 2.3 (1.14) | -1.9 (1.08)
  Mental Health, Year 1 | 2.7 (0.98) | -2.1 (0.96)
  Mental Health, Year 2 | 2.0 (1.07) | -0.4 (1.02)
  Physical Function, Year 1 | 3.5 (1.1) | -2.1 (1.1)
  Physical Function, Year 2 | -2.5 (1.33) | -2.5 (1.27)
  Physical Role, Year 1 | 2.6 (2.23) | -5.5 (2.20)
  Physical Role, Year 2 | -2.3 (2.59) | -7.3 (2.47)
  Social Function, Year 1 | 1.8 (1.23) | -3.0 (1.21)
  Social Function, Year 2 | -0.1 (1.44) | -3.0 (1.37)
  Vitality Function, Year 1 | 3.9 (0.97) | -0.6 (0.95)
  Vitality Function, Year 2 | 2.8 (1.10) | -1.0 (1.05)
  Bodily Pain, Year 1 | -0.2 (1.37) | -2.1 (1.35)
  Bodily Pain, Year 2 | -2.0 (1.53) | -1.2 (1.46)
  Emotional Role, Year 1 | 0.4 (2.17) | -4.3 (2.14)
  Emotional Role, Year 2 | -0.1 (2.51) | -2.2 (2.42)
Statistical Analysis 1: Comparison: Early Epoetin Beta Therapy vs Late Epoetin Beta Therapy; Mean Change from Baseline in the Score of General health scale of Quality of life for Year 1; Test type: Superiority or Other; p = 0.0029, ANCOVA
Statistical Analysis 2: Comparison: Early Epoetin Beta Therapy vs Late Epoetin Beta Therapy; Mean Change from Baseline in the Score of General health scale of Quality of life for Year 2; Test type: Superiority or Other; p = 0.0081, ANCOVA
Statistical Analysis 3: Comparison: Early Epoetin Beta Therapy vs Late Epoetin Beta Therapy; Mean Change from Baseline in the Score of Mental health scale of Quality of life for Year 1; Test type: Superiority or Other; p = 0.0005, ANCOVA
Statistical Analysis 4: Comparison: Early Epoetin Beta Therapy vs Late Epoetin Beta Therapy; Mean Change from Baseline in the Score of Mental Health scale of Quality of life for Year 2; Test type: Superiority or Other; p = 0.0965, ANCOVA
Statistical Analysis 5: Comparison: Early Epoetin Beta Therapy vs Late Epoetin Beta Therapy; Mean Change from Baseline in the Score of Physical function scale of Quality of life for Year 1; Test type: Superiority or Other; p = 0.0004, ANCOVA
Statistical Analysis 6: Comparison: Early Epoetin Beta Therapy vs Late Epoetin Beta Therapy; Mean Change from Baseline in the Score of Physical function scale of Quality of life for Year 2; Test type: Superiority or Other; p = 0.9864, ANCOVA
Statistical Analysis 7: Comparison: Early Epoetin Beta Therapy vs Late Epoetin Beta Therapy; Mean Change from Baseline in the Score of Physical Role scale of Quality of life for Year 1; Test type: Superiority or Other; p = 0.0097, ANCOVA
Statistical Analysis 8: Comparison: Early Epoetin Beta Therapy vs Late Epoetin Beta Therapy; Mean Change from Baseline in the Score of Physical Role scale of Quality of life for Year 2; Test type: Superiority or Other; p = 0.1670, ANCOVA
Statistical Analysis 9: Comparison: Early Epoetin Beta Therapy vs Late Epoetin Beta Therapy; Mean Change from Baseline in the Score of Social function scale of Quality of life for Year 1; Test type: Superiority or Other; p = 0.0058, ANCOVA
Statistical Analysis 10: Comparison: Early Epoetin Beta Therapy vs Late Epoetin Beta Therapy; Mean Change from Baseline in the Score of Social function scale of Quality of life for Year 2; Test type: Superiority or Other; p = 0.1455, ANCOVA
Statistical Analysis 11: Comparison: Early Epoetin Beta Therapy vs Late Epoetin Beta Therapy; Mean Change from Baseline in the Score of Vitality function scale of Quality of life for Year 1; Test type: Superiority or Other; p = 0.0009, ANCOVA
Statistical Analysis 12: Comparison: Early Epoetin Beta Therapy vs Late Epoetin Beta Therapy; Mean Change from Baseline in the Score of Vitality function scale of Quality of life for Year 2; Test type: Superiority or Other; p = 0.0123, ANCOVA
Statistical Analysis 13: Comparison: Early Epoetin Beta Therapy vs Late Epoetin Beta Therapy; Mean Change from Baseline in the Score of Bodily pain scale of Quality of life for Year 1; Test type: Superiority or Other; p = 0.3155, ANCOVA
Statistical Analysis 14: Comparison: Early Epoetin Beta Therapy vs Late Epoetin Beta Therapy; Mean Change from Baseline in the Score of Bodily pain scale of Quality of life for Year 2; Test type: Superiority or Other; p = 0.7076, ANCOVA
Statistical Analysis 15: Comparison: Early Epoetin Beta Therapy vs Late Epoetin Beta Therapy; Mean Change from Baseline in the Score of Emotional role scale of Quality of life for Year 1; Test type: Superiority or Other; p = 0.1291, ANCOVA
Statistical Analysis 16: Comparison: Early Epoetin Beta Therapy vs Late Epoetin Beta Therapy; Mean Change from Baseline in the Score of Emotional role scale of Quality of life for Year 2; Test type: Superiority or Other; p = 0.5528, ANCOVA

17. Secondary Outcome: Number of Participants on Blood Pressure/Anti-Hypertensive Treatment According to Class Of Drugs
Description: Anti-hypertensive is defined as class of drugs that are used to treat hypertension. Numbers (No.) of participants treated with at least one hypertensive medication/Treatment (Tt) according to class of drugs were reported.
Time Frame: Up to 4 years
Population: The safety analysis population included all participants who were randomized and who had received a safety follow-up whether or not they had received epoetin beta treatment.
Measure: Number; unit: participants
Arm/Group | Early Epoetin Beta Therapy | Late Epoetin Beta Therapy
Number analyzed (Participants) | 300 | 302
participants
  No. of participants with at least one Tt | 287 | 282
  Calcium Channel Blocking Agents | 201 | 204
  Loop Diuretics | 183 | 180
  Angiotensin-Converting Enzyme Inhibitors | 158 | 153
  Beta-Adrenoceptor Blocking Agents | 169 | 136
  Angiotensin-II Receptor Antagonists | 89 | 96
  Alpha-Adrenoreceptor Antagonists | 87 | 73
  Antihypertensive Agents | 55 | 52
  Thiazide And Related Diuretics | 44 | 40
  Antianginal Agents | 6 | 5
  Potassium Sparing Diuretics | 4 | 7
  Aldosterone Antagonists | 2 | 5
  Cardiac Glycosides | 1 | 1
  Diuretics | 2 | 0
  Supplements | 1 | 1
  Calcium Compounds And Regulators | 0 | 1
  Miscellaneous Drugs | 0 | 1
  Tricyclic Antidepressants | 1 | 0

18. Secondary Outcome: Number of Participants With Marked Laboratory Abnormalities
Description: Marked abnormality of laboratory parameters is defined as the value which is outside the defined reference range of that respective parameter. Values above and below the given reference range were determined as High or Low range values of the laboratory parameter. Roche's standard reference ranges for laboratory test parameters were used for the analysis. The laboratory parameters with marked abnormality are platelets (reference range is 150-350 10^9 cells/liter [L]), creatinine (reference range is 0-133 micromole per liter), albumin (reference range is 35.0-55 g/L), phosphate (reference range is 0.84-1.45 millimole per liter [mmol /L]) and potassium (reference range is 3.4-4.8 mmol /L).
Time Frame: Baseline, every 3 months up to 4 years
Population: The safety analysis population included all participants who were randomized and who had received a safety follow-up whether or not they had received epoetin beta treatment. The ''n" represents the number of participants assessed for each laboratory parameter.
Measure: Number; unit: participants
Arm/Group | Early Epoetin Beta Therapy | Late Epoetin Beta Therapy
Number analyzed (Participants) | 206 | 208
participants
  Platelets - High; n = 206, 208 | 5 | 0
  Platelets - Low; n = 206, 208 | 13 | 15
  Creatinine - High; n = 206, 208 | 140 | 128
  Albumin - Low; n = 201, 205 | 6 | 9
  Phosphate - High; n = 206, 208 | 164 | 150
  Phosphate - Low; n = 206, 208 | 22 | 23
  Potassium - High; n = 206, 208 | 47 | 46
  Potassium - Low; n = 206, 208 | 4 | 6

ADVERSE EVENTS:
Time Frame: Up to 4 years
Description: An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Arm/Group | Early Epoetin Beta Therapy | Late Epoetin Beta Therapy
Serious Adverse Events (participants affected / at risk) | 158/300 | 145/302
Other Adverse Events (participants affected / at risk) | 243/300 | 228/302
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Early Epoetin Beta Therapy (N=300) | Late Epoetin Beta Therapy (N=302)
Pneumonia (Infections and infestations) | 9 | 9
Urinary Tract Infection (Infections and infestations) | 4 | 8
Sepsis (Infections and infestations) | 6 | 3
Gastroenteritis (Infections and infestations) | 2 | 4
Renal Cyst Infection (Infections and infestations) | 1 | 4
Appendicitis (Infections and infestations) | 2 | 2
Upper Respiratory Tract Infection (Infections and infestations) | 2 | 2
Erysipelas (Infections and infestations) | 2 | 1
Respiratory Tract Infection (Infections and infestations) | 1 | 2
Abscess Limb (Infections and infestations) | 0 | 2
Bacteraemia (Infections and infestations) | 2 | 0
Bronchopneumonia (Infections and infestations) | 1 | 1
Catheter Related Infection (Infections and infestations) | 2 | 0
Catheter Site Infection (Infections and infestations) | 1 | 1
Diverticulitis (Infections and infestations) | 1 | 1
Herpes Zoster (Infections and infestations) | 1 | 1
Pyelonephritis (Infections and infestations) | 2 | 0
Pyelonephritis Acute (Infections and infestations) | 1 | 1
Sepsis Syndrome (Infections and infestations) | 2 | 0
Bronchitis Acute (Infections and infestations) | 0 | 1
Catheter Sepsis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Cholecystitis Infective (Infections and infestations) | 1 | 0
Clostridial Infection (Infections and infestations) | 1 | 0
Epidemic Nephropathy (Infections and infestations) | 0 | 1
Escherichia Sepsis (Infections and infestations) | 1 | 0
Fungal Peritonitis (Infections and infestations) | 0 | 1
Hepatic Cyst Infection (Infections and infestations) | 1 | 0
Hepatitis C (Infections and infestations) | 1 | 0
Infected Skin Ulcer (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 1 | 0
Kidney Infection (Infections and infestations) | 1 | 0
Localised Infection (Infections and infestations) | 0 | 2
Lower Respiratory Tract Infection (Infections and infestations) | 1 | 0
Lung Infection (Infections and infestations) | 0 | 1
Pneumonia Fungal (Infections and infestations) | 1 | 0
Sialoadenitis (Infections and infestations) | 1 | 0
Staphylococcal Sepsis (Infections and infestations) | 0 | 1
Streptococcal Sepsis (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0
Wound Infection (Infections and infestations) | 0 | 1
Arrhythmia (Cardiac disorders) | 16 | 14
Cardiac Failure Acute (Cardiac disorders) | 11 | 19
Myocardial Infarction (Cardiac disorders) | 13 | 14
Angina Pectoris (Cardiac disorders) | 11 | 4
Cardiac Arrest (Cardiac disorders) | 2 | 0
Cardiac Failure Chronic (Cardiac disorders) | 0 | 1
Cardiac Failure Congestive (Cardiac disorders) | 0 | 1
Cardiopulmonary Failure (Cardiac disorders) | 1 | 0
Coronary Artery Occlusion (Cardiac disorders) | 1 | 0
Coronary Artery Stenosis (Cardiac disorders) | 1 | 1
Myocarditis (Cardiac disorders) | 1 | 0
Pericardial Effusion (Cardiac disorders) | 0 | 1
Renal Failure (Renal and urinary disorders) | 17 | 12
Renal Impairment (Renal and urinary disorders) | 5 | 9
Renal Failure Chronic (Renal and urinary disorders) | 7 | 6
Azotaemia (Renal and urinary disorders) | 5 | 1
Haematuria (Renal and urinary disorders) | 4 | 1
Urinary Retention (Renal and urinary disorders) | 1 | 3
Hydronephrosis (Renal and urinary disorders) | 0 | 2
Renal Cyst Ruptured (Renal and urinary disorders) | 1 | 1
Renal Failure Acute (Renal and urinary disorders) | 1 | 1
Renal Haemorrhage (Renal and urinary disorders) | 1 | 1
Calculus Ureteric (Renal and urinary disorders) | 1 | 0
Glomerulonephritis (Renal and urinary disorders) | 0 | 1
Haemorrhage Urinary Tract (Renal and urinary disorders) | 1 | 0
Hypertensive Nephropathy (Renal and urinary disorders) | 0 | 1
Nephritis Interstitial (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Renal Artery Stenosis (Renal and urinary disorders) | 0 | 1
Urinary Bladder Polyp (Renal and urinary disorders) | 1 | 0
Peritonitis (Gastrointestinal disorders) | 4 | 3
Abdominal Pain (Gastrointestinal disorders) | 0 | 5
Vomiting (Gastrointestinal disorders) | 1 | 4
Diarrhoea (Gastrointestinal disorders) | 2 | 2
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 3 | 1
Pancreatitis Acute (Gastrointestinal disorders) | 1 | 3
Gastritis (Gastrointestinal disorders) | 3 | 0
Intestinal Ischaemia (Gastrointestinal disorders) | 1 | 2
Constipation (Gastrointestinal disorders) | 2 | 0
Diverticulum Intestinal (Gastrointestinal disorders) | 2 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 2
Ileus (Gastrointestinal disorders) | 1 | 1
Inguinal Hernia (Gastrointestinal disorders) | 2 | 0
Abdominal Haematoma (Gastrointestinal disorders) | 1 | 0
Abdominal Hernia (Gastrointestinal disorders) | 1 | 0
Abdominal Symptom (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Colitis Ulcerative (Gastrointestinal disorders) | 0 | 1
Colonic Polyp (Gastrointestinal disorders) | 1 | 0
Diverticular Perforation (Gastrointestinal disorders) | 0 | 1
Duodenal Ulcer (Gastrointestinal disorders) | 1 | 0
Duodenitis Haemorrhagic (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0
Erosive Duodenitis (Gastrointestinal disorders) | 1 | 0
Gastric Haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastric Ulcer (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0
Ileus Paralytic (Gastrointestinal disorders) | 0 | 1
Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis Chronic (Gastrointestinal disorders) | 0 | 1
Peptic Ulcer (Gastrointestinal disorders) | 0 | 1
Reflux Oesophagitis (Gastrointestinal disorders) | 1 | 0
Arteriovenous Fistula Thrombosis (Injury, poisoning and procedural complications) | 0 | 4
Hip Fracture (Injury, poisoning and procedural complications) | 1 | 3
Arteriovenous Fistula Site Complication (Injury, poisoning and procedural complications) | 3 | 0
Complications Of Transplanted Kidney (Injury, poisoning and procedural complications) | 1 | 1
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 2 | 0
Head Injury (Injury, poisoning and procedural complications) | 1 | 1
Humerus Fracture (Injury, poisoning and procedural complications) | 1 | 1
Acetabulum Fracture (Injury, poisoning and procedural complications) | 0 | 1
Arterial Injury (Injury, poisoning and procedural complications) | 1 | 0
Arteriovenous Fistula Site Haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Cardiac Pacemaker Malfunction (Injury, poisoning and procedural complications) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Eye Injury (Injury, poisoning and procedural complications) | 1 | 0
Femur Fracture (Injury, poisoning and procedural complications) | 0 | 1
Injury (Injury, poisoning and procedural complications) | 1 | 0
Joint Injury (Injury, poisoning and procedural complications) | 1 | 0
Medical Device Complication (Injury, poisoning and procedural complications) | 1 | 0
Medication Error (Injury, poisoning and procedural complications) | 1 | 0
Multiple Fractures (Injury, poisoning and procedural complications) | 0 | 1
Open Wound (Injury, poisoning and procedural complications) | 1 | 0
Post Procedural Haematoma (Injury, poisoning and procedural complications) | 1 | 0
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Postoperative Hernia (Injury, poisoning and procedural complications) | 0 | 1
Procedural Complication (Injury, poisoning and procedural complications) | 1 | 0
Renal Haematoma (Injury, poisoning and procedural complications) | 1 | 0
Shunt Thrombosis (Injury, poisoning and procedural complications) | 1 | 0
Subdural Haematoma (Injury, poisoning and procedural complications) | 1 | 0
Subdural Haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Vascular Access Complication (Injury, poisoning and procedural complications) | 0 | 1
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Renal Cell Carcinoma Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Bladder Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cervix Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gallbladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gammopathy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Laryngeal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases To Liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Parathyroid Tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostatic Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tongue Neoplasm Malignant Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Lung Disorder (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Chronic Obstructive Airways Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Laryngeal Dysplasia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Vocal Cord Polyp (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 6 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 3 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 2
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 2 | 1
Fluid Overload (Metabolism and nutrition disorders) | 3 | 0
Fluid Retention (Metabolism and nutrition disorders) | 2 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 3
Metabolic Acidosis (Metabolism and nutrition disorders) | 2 | 1
Diabetes Mellitus (Metabolism and nutrition disorders) | 1 | 1
Diabetic Foot (Metabolism and nutrition disorders) | 0 | 1
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Electrolyte Imbalance (Metabolism and nutrition disorders) | 0 | 1
Gout (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Cerebrovascular Accident (Nervous system disorders) | 7 | 5
Syncope (Nervous system disorders) | 1 | 3
Headache (Nervous system disorders) | 2 | 1
Diabetic Neuropathy (Nervous system disorders) | 2 | 0
Dizziness (Nervous system disorders) | 1 | 1
Transient Ischaemic Attack (Nervous system disorders) | 2 | 0
Carotid Artery Stenosis (Nervous system disorders) | 0 | 1
Carpal Tunnel Syndrome (Nervous system disorders) | 1 | 0
Cervical Root Pain (Nervous system disorders) | 0 | 1
Cervicobrachial Syndrome (Nervous system disorders) | 0 | 1
Dementia Alzheimer's Type (Nervous system disorders) | 0 | 1
Diabetic Hyperglycaemic Coma (Nervous system disorders) | 1 | 0
Disturbance In Attention (Nervous system disorders) | 1 | 0
Dizziness Postural (Nervous system disorders) | 0 | 1
Hypersomnia (Nervous system disorders) | 1 | 0
Hypertonia (Nervous system disorders) | 1 | 0
Loss Of Consciousness (Nervous system disorders) | 0 | 1
Neuralgia (Nervous system disorders) | 0 | 1
Uraemic Encephalopathy (Nervous system disorders) | 1 | 0
Pyrexia (General disorders) | 3 | 4
Sudden Death (General disorders) | 4 | 2
Oedema Peripheral (General disorders) | 3 | 1
Chest Pain (General disorders) | 3 | 0
Asthenia (General disorders) | 1 | 1
Catheter Related Complication (General disorders) | 1 | 1
General Physical Health Deterioration (General disorders) | 0 | 2
Oedema (General disorders) | 1 | 1
Adverse Drug Reaction (General disorders) | 0 | 1
Catheter Site Inflammation (General disorders) | 1 | 0
Chills (General disorders) | 1 | 0
Fatigue (General disorders) | 0 | 1
Heparin-Induced Thrombocytopenia (General disorders) | 1 | 0
Injection Site Thrombosis (General disorders) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 4 | 0
Localised Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Gouty Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint Swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Cholecystitis Acute (Hepatobiliary disorders) | 2 | 3
Cholelithiasis (Hepatobiliary disorders) | 1 | 2
Cholecystitis (Hepatobiliary disorders) | 0 | 2
Cholestasis Of Pregnancy (Hepatobiliary disorders) | 1 | 0
Hepatic Cyst (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 1
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 1 | 0
Epididymitis (Reproductive system and breast disorders) | 1 | 0
Ovarian Cyst (Reproductive system and breast disorders) | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 1 | 0
Uterine Prolapse (Reproductive system and breast disorders) | 0 | 1
Nephrectomy (Surgical and medical procedures) | 2 | 1
Insertion Of Ambulatory Peritoneal Catheter (Surgical and medical procedures) | 1 | 1
Arteriovenous Fistula Operation (Surgical and medical procedures) | 0 | 1
Cataract Operation (Surgical and medical procedures) | 0 | 1
Catheter Placement (Surgical and medical procedures) | 1 | 0
Eye Operation (Surgical and medical procedures) | 1 | 0
Knee Arthroplasty (Surgical and medical procedures) | 1 | 0
Peritoneal Dialysis (Surgical and medical procedures) | 1 | 0
Rehabilitation Therapy (Surgical and medical procedures) | 1 | 0
Renal Transplant (Surgical and medical procedures) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 3 | 6
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Nephrogenic Anaemia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Blood Pressure Increased (Investigations) | 3 | 0
Biopsy Liver (Investigations) | 1 | 0
Blood Creatine Phosphokinase Increased (Investigations) | 0 | 1
Transaminases Increased (Investigations) | 0 | 1
Urine Cytology Abnormal (Investigations) | 1 | 0
Weight Decreased (Investigations) | 1 | 0
Weight Increased (Investigations) | 0 | 1
Skin Ulcer (Skin and subcutaneous tissue disorders) | 0 | 3
Angioneurotic Oedema (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Retinal Detachment (Eye disorders) | 1 | 1
Cataract (Eye disorders) | 0 | 1
Glaucoma (Eye disorders) | 1 | 0
Ocular Hypertension (Eye disorders) | 0 | 1
Strabismus (Eye disorders) | 0 | 1
Vitreous Haemorrhage (Eye disorders) | 0 | 1
Hyperparathyroidism (Endocrine disorders) | 0 | 2
Hyperparathyroidism Secondary (Endocrine disorders) | 2 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 1
Confusional State (Psychiatric disorders) | 2 | 0
Amnestic Disorder (Psychiatric disorders) | 1 | 0
Disorientation (Psychiatric disorders) | 1 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 2 | 1
Premature Labour (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Congenital Cystic Kidney Disease (Congenital, familial and genetic disorders) | 1 | 0
Polycystic Liver Disease (Congenital, familial and genetic disorders) | 0 | 1
Amyloidosis (Immune system disorders) | 1 | 0
Kidney Transplant Rejection (Immune system disorders) | 1 | 0
Vestibular Neuronitis (Ear and labyrinth disorders) | 1 | 0
Peripheral Vascular Disorder (Vascular disorders) | 12 | 7
Hypotension (Vascular disorders) | 2 | 2
Deep Vein Thrombosis (Vascular disorders) | 1 | 2
Arterial Stenosis (Vascular disorders) | 2 | 0
Hypertension (Vascular disorders) | 0 | 2
Hypertensive Crisis (Vascular disorders) | 2 | 0
Lymphocele (Vascular disorders) | 1 | 1
Phlebitis (Vascular disorders) | 2 | 0
Aneurysm Arteriovenous (Vascular disorders) | 1 | 0
Aortic Aneurysm (Vascular disorders) | 1 | 0
Arteriosclerosis (Vascular disorders) | 0 | 1
Arteriovenous Fistula, Acquired (Vascular disorders) | 0 | 1
Circulatory Collapse (Vascular disorders) | 1 | 0
Malignant Hypertension (Vascular disorders) | 1 | 0
Orthostatic Hypotension (Vascular disorders) | 1 | 0
Subclavian Artery Aneurysm (Vascular disorders) | 1 | 0
Thrombophlebitis (Vascular disorders) | 1 | 0
Venous Thrombosis Limb (Vascular disorders) | 0 | 1
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Early Epoetin Beta Therapy (N=300) | Late Epoetin Beta Therapy (N=302)
Renal Failure (Renal and urinary disorders) | 93 | 87
Renal Failure Chronic (Renal and urinary disorders) | 33 | 46
Renal Impairment (Renal and urinary disorders) | 27 | 23
Upper respiratory tract infection (Infections and infestations) | 16 | 28
Urinary tract infection (Infections and infestations) | 26 | 29
Nasopharyngitis (Infections and infestations) | 24 | 23
Influenza (Infections and infestations) | 26 | 12
Bronchitis (Infections and infestations) | 12 | 16
Bronchitis Acute (Infections and infestations) | 15 | 6
Hypertension (Vascular disorders) | 89 | 58
Hypotension (Vascular disorders) | 13 | 16
Diarrhoea (Gastrointestinal disorders) | 24 | 25
Constipation (Gastrointestinal disorders) | 22 | 19
Nausea (Gastrointestinal disorders) | 15 | 14
Vomiting (Gastrointestinal disorders) | 15 | 12
Back pain (Musculoskeletal and connective tissue disorders) | 22 | 33
Arthralgia (Musculoskeletal and connective tissue disorders) | 21 | 19
Pain in extremity (Musculoskeletal and connective tissue disorders) | 18 | 16
Muscle cramp (Musculoskeletal and connective tissue disorders) | 9 | 16
Hyperkalaemia (Metabolism and nutrition disorders) | 28 | 30
Hyperphosphataemia (Metabolism and nutrition disorders) | 27 | 22
Gout (Metabolism and nutrition disorders) | 15 | 16
Oedema Peripheral (General disorders) | 20 | 11
Asthenia (General disorders) | 16 | 17
Fatigue (General disorders) | 14 | 17
Headache (Nervous system disorders) | 30 | 15
Dizziness (Nervous system disorders) | 18 | 13
Pruritis (Skin and subcutaneous tissue disorders) | 27 | 18
Cough (Respiratory, thoracic and mediastinal disorders) | 20 | 16
Insomnia (Psychiatric disorders) | 12 | 23
Blood Pressure Increased (Investigations) | 19 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.